CLINICAL TRIAL: NCT00064961
Title: Obesity Prevention After Smoking Cessation in Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG0004
Record Dates: First submitted 2003-07-16; First posted 2003-07-17 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Obesity; Menopause
Keywords: Smoking Cessation
MeSH Terms: conditions — Obesity; Smoking Cessation

INTERVENTIONS:
Behavioral: Individualized dietary-control and exercise program
Behavioral: Weight-management and smoking cessation maintenance
Behavioral: Smoking Cessation program

SUMMARY:
This study addresses the high risk of weight gain associated with smoking cessation in women. The obesity prevention pilot study is designed for the primary prevention of weight gain that can lead to overweight in normal-weight women, that can progress to obesity in women who are already overweight, and for the prevention of additional weight gain in obese women with BMI greater than or equal to 30.0. Fat and other macronutrient intake, specifically, sugar, complex carbohydrates, and protein, are analyzed as a target for individually tailored, weight control intervention following smoking cessation in Caucasian and African American women.

DETAILED DESCRIPTION:
Middle-aged women, especially African Americans, who quit smoking are at high risk for weight gain, overweight, and obesity. Postcessation weight gain has been attributed to increased food intake, which in turn, has been ascribed to a selective increase in high-sugar and other high-carbohydrate foods with a high-fat content. This study compares the relative effectiveness, for postmenopausal Caucasian and African American women, of following an empirically validated smoking cessation program with either 1) a group cessation maintenance program with standard exercise advice and food pyramid instructions for healthy eating or 2) an individually tailored, dietary-control, exercise, weight-management and cessation-maintenance program. Effectiveness is assessed by weight change from baseline to postcessation months 6, 12, and 20.

The second aim is to assess overall fat and other specific macronutrient intake (sugar, complex carbohydrates, and protein) and total caloric intake with the use of a novel macronutrient self-selection paradigm in Caucasian and African-American postmenopausal women at baseline prior to smoking cessation, after being abstinent for one week, and again at 6, 12, and 20 months postcessation.

The third aim is to assess whether there is differential responsiveness on the above measures in postmenopausal Caucasian vs. African-American women.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 45 - 59 at time of enrollment
* African-American or Caucasian; able to confirm racial heritage of past two generations in family
* Postmenopausal
* Smokers (more than 10 cigarettes per day for 1 year or more)
* Written physician approval to participate in program and medical clearance that use of over-the-counter nicotine replacement is not contraindicated based on patient's medical status

Exclusion Criteria

* Men
* Age below 45 or above 59
* Nonsmokers
* Currently in a standardized weight-reduction program or taking medications for weight loss
* History or presence of significant psychiatric illness (e.g., eating disorders, psychosis, psychoactive substance abuse, major depression)
* History of presence of severe physical illness (e.g., renal failure, hepatic failure, cancer, immunological disease)
* Unable to complete long-term study commitment, including anticipating moving out of study area prior to completion of the study
* Unable to confirm racial heritage of past two generations in family.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2000-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Pirie PL, McBride CM, Hellerstedt W, Jeffery RW, Hatsukami D, Allen S, Lando H. Smoking cessation in women concerned about weight. Am J Public Health. 1992 Sep;82(9):1238-43. doi: 10.2105/ajph.82.9.1238. PMID 1503165
- [Background] Williamson DF, Madans J, Anda RF, Kleinman JC, Giovino GA, Byers T. Smoking cessation and severity of weight gain in a national cohort. N Engl J Med. 1991 Mar 14;324(11):739-45. doi: 10.1056/NEJM199103143241106. PMID 1997840
- [Background] Hall SM, Tunstall CD, Vila KL, Duffy J. Weight gain prevention and smoking cessation: cautionary findings. Am J Public Health. 1992 Jun;82(6):799-803. doi: 10.2105/ajph.82.6.799. PMID 1585959
- [Background] Heymsfield SB, Gallagher D, Poehlman ET, Wolper C, Nonas K, Nelson D, Wang ZM. Menopausal changes in body composition and energy expenditure. Exp Gerontol. 1994 May-Aug;29(3-4):377-89. doi: 10.1016/0531-5565(94)90018-3. PMID 7925757
- [Background] Geiselman PJ, Anderson AM, Dowdy ML, West DB, Redmann SM, Smith SR. Reliability and validity of a macronutrient self-selection paradigm and a food preference questionnaire. Physiol Behav. 1998 Mar;63(5):919-28. doi: 10.1016/s0031-9384(97)00542-8. PMID 9618017